CLINICAL TRIAL: NCT03425643
Title: A Phase III, Randomized, Double-blind Trial of Platinum Doublet Chemotherapy +/-Pembrolizumab (MK-3475) as Neoadjuvant/Adjuvant Therapy for Participants With Resectable Stage II, IIIA, and Resectable IIIB (T3-4N2) Non-small Cell Lung Cancer (NSCLC) (KEYNOTE-671)
Brief Title: Efficacy and Safety of Pembrolizumab (MK-3475) With Platinum Doublet Chemotherapy as Neoadjuvant/Adjuvant Therapy for Participants With Resectable Stage II, IIIA, and Resectable IIIB (T3-4N2) Non-small Cell Lung Cancer (MK-3475-671/KEYNOTE-671)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-671; MK-3475-671 (Other: MSD); 183970 (Other: JAPIC-CTI); 2017-001832-21 (EudraCT Number)
Record Dates: First submitted 2018-02-02; First posted 2018-02-07 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Cisplatin; Gemcitabine; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NAC + Neoadjuvant/Adjuvant Pembrolizumab (Experimental): Neoadjuvant: Prior to surgery, participants receive up to 4 cycles (cycle length: 3 weeks) of pembrolizumab [200 mg, intravenous (IV); given on cycle day 1] in combination with platinum doublet neoadjuvant chemotherapy (NAC), consisting of cisplatin [75 mg/m^2, IV; given on cycle day 1] and either Gemcitabine [1000 mg/m^2, IV; given on cycle days 1 and 8] or Pemetrexed [500 mg/m^2, IV; given on cycle day 1].
  Adjuvant: 4-12 weeks following surgery, participants receive 13 cycles (cycle length: 3 weeks) of pembrolizumab [200 mg, IV; given on cycle day 1].
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: Gemcitabine; Drug: Pemetrexed
- NAC + Neoadjuvant/Adjuvant Placebo (Placebo Comparator): Neoadjuvant: Prior to surgery, participants receive up to 4 cycles (cycle length: 3 weeks) of placebo [normal saline, IV; given on cycle day 1] in combination with platinum doublet NAC, consisting of cisplatin [75 mg/m^2, IV; given on cycle day 1] and either Gemcitabine [1000 mg/m^2, IV; given on cycle days 1 and 8] or Pemetrexed [500 mg/m^2, IV; given on cycle day 1].
  Adjuvant: 4-12 weeks following surgery, participants receive 13 cycles (cycle length: 3 weeks) of placebo [normal saline, IV; given on cycle day 1].
  Interventions: Drug: Placebo; Drug: Cisplatin; Drug: Gemcitabine; Drug: Pemetrexed

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg by IV infusion every 3 weeks (Q3W), given on cycle day 1.
  Other Names: KEYTRUDA®; MK-3475
  Arms: NAC + Neoadjuvant/Adjuvant Pembrolizumab
Drug: Placebo — Normal saline by IV infusion Q3W, given on cycle day 1.
  Arms: NAC + Neoadjuvant/Adjuvant Placebo
Drug: Cisplatin — 75 mg/m^2 by IV infusion Q3W, given on cycle day 1.
  Other Names: PLATINOL®
Drug: Gemcitabine — 1000 mg/m^2 by IV infusion Q3W, given on cycle days 1 and 8. Given only to participants with squamous NSCLC.
  Other Names: GEMZAR®
Drug: Pemetrexed — 500 mg/m^2 by IV infusion Q3W, given on cycle day 1. Given only to participants with nonsquamous NSCLC.
  Other Names: Alimta®

SUMMARY:
This trial will evaluate the safety and efficacy of pembrolizumab (MK-3475) in combination with platinum doublet neoadjuvant chemotherapy (NAC) before surgery [neoadjuvant phase], followed by pembrolizumab alone after surgery [adjuvant phase] in participants with resectable stage II, IIIA, and resectable IIIB (T3-4N2) non-small cell lung cancer (NSCLC). The primary hypotheses of this study are that neoadjuvant pembrolizumab (vs. placebo) in combination with NAC, followed by surgery and adjuvant pembrolizumab (vs. placebo) will improve: 1) event free survival (EFS) by biopsy assessed by local pathologist or by investigator-assessed imaging using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1); and 2) overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Have previously untreated and pathologically confirmed resectable Stage II, IIIA, or IIIB (N2) NSCLC.
* If male, must agree to use contraception or practice abstinence as well as refrain from donating sperm during the treatment period and for the time needed to eliminate each study intervention after the last dose of study intervention.
* If female, may participate if not pregnant or breastfeeding, and at least one of the following conditions apply: 1) not a woman of childbearing potential (WOCBP); or 2) a WOCBP who agrees to follow contraceptive guidance during the treatment period and for the time needed to eliminate each study intervention after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) to others or freeze/store for her own use for the purpose of reproduction during this period.
* Have available formalin-fixed paraffin embedded (FFPE) tumor tissue sample blocks for submission. If blocks are not available, have unstained slides for submission for central programmed death-ligand 1 (PD-L1) testing.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 10 days of randomization.
* Have adequate organ function.

Exclusion Criteria:

* Has one of the following tumor locations/types:1) NSCLC involving the superior sulcus; 2) Large cell neuro-endocrine cancer (LCNEC); or 3) Sarcomatoid tumor.
* Has a history of (non-infectious) pneumonitis /interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease that requires steroids.
* Has an active infection requiring systemic therapy.
* Has had an allogenic tissue/sold organ transplant.
* Has a known severe hypersensitivity (≥ Grade 3) to pembrolizumab, its active substance and/or any of its excipients.
* Has a known severe hypersensitivity (≥ Grade 3) to any of the study chemotherapy agents and/or to any of their excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of Hepatitis B or Hepatitis C.
* Has a known history of active tuberculosis.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate.
* Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the trial.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor.
* Has received prior systemic anti-cancer therapy including investigational agents for the current malignancy prior to randomization/allocation.
* Has received prior radiotherapy within 2 weeks of start of trial treatment.
* Has received a live vaccine within 30 days prior to the first dose of trial drug.
* Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of trial treatment.
* Has a diagnosis of immunodeficiency or is receiving either systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of trial drug.
* Has a known additional malignancy that is progressing or requires active treatment within the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 797 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2026-06-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (227):
- United States (51):
  - Banner MD Anderson Cancer Center ( Site 0028), Gilbert, Arizona
  - Western Regional Medical Center, Inc. ( Site 0050), Goodyear, Arizona
  - University of Arizona Cancer Center - Dignity Health ( Site 0062), Phoenix, Arizona
  - University of Arizona Cancer Center ( Site 0012), Tucson, Arizona
  - Pacific Cancer Medical Center, Inc. ( Site 0004), Anaheim, California
  - Providence Saint Joseph Medical Center ( Site 0061), Burbank, California
  - Pacific Cancer Care ( Site 0035), Monterey, California
  - John Wayne Cancer Institute ( Site 0049), Santa Monica, California
  - St Joseph Heritage Healthcare ( Site 0040), Santa Rosa, California
  - Stanford University, Stanford Cancer Center ( Site 0046), Stanford, California
  - Hartford Hospital ( Site 0069), Hartford, Connecticut
  - Helen F. Graham Cancer Center & Research Institute ( Site 0015), Newark, Delaware
  - Mayo Clinic Jacksonville ( Site 0022), Jacksonville, Florida
  - Miami Cancer Institute-Baptist Hospital ( Site 0068), Miami, Florida
  - Southeastern Regional Medical Center ( Site 0051), Newnan, Georgia
  - Northwest Oncology and Hematology ( Site 0001), Elk Grove Village, Illinois
  - Ingalls Memorial Hospital ( Site 0044), Harvey, Illinois
  - PPG-Oncology ( Site 0043), Fort Wayne, Indiana
  - University of Iowa Hospital and Clinics ( Site 0010), Iowa City, Iowa
  - Ashland-Bellefonte Cancer Center ( Site 0021), Ashland, Kentucky
  - Harry & Jeanette Weinberg Cancer Institute ( Site 0081), Baltimore, Maryland
  - Boston Medical Center ( Site 0057), Boston, Massachusetts
  - UMass Memorial Medical Center ( Site 0030), Worcester, Massachusetts
  - Henry Ford Health System ( Site 0031), Detroit, Michigan
  - Herbert Herman Cancer Center, Sparrow Hospital ( Site 0034), Lansing, Michigan
  - Mayo Clinic ( Site 0026), Rochester, Minnesota
  - St. Vincent Healthcare Frontier Cancer Center ( Site 0005), Billings, Montana
  - University of Nebraska Medical Center ( Site 0047), Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center Basking Ridge ( Site 0074), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center- Monmouth ( Site 0077), Middletown, New Jersey
  - MSKCC-Bergen ( Site 0075), Montvale, New Jersey
  - St. Peter's Hospital Cancer Care Center ( Site 0039), Albany, New York
  - Memorial Sloan-Kettering Cancer Center at Commack ( Site 0076), Commack, New York
  - Memorial Sloan Kettering Cancer Center Westchester ( Site 0079), Harrison, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0060), New York, New York
  - Stony Brook University Medical Center - Cancer Center ( Site 0019), Stony Brook, New York
  - Montefiore Einstein Center ( Site 0016), The Bronx, New York
  - Memorial Sloan Kettering Cancer Center - Nassau ( Site 0078), Uniondale, New York
  - White Plains Hospital Center for Cancer Care ( Site 0007), White Plains, New York
  - Southwestern Regional Medical Center, Inc. ( Site 0054), Tulsa, Oklahoma
  - OHSU Center for Health & Healing ( Site 1006), Portland, Oregon
  - UPMC Pinnacle Health System - East Location ( Site 0063), Harrisburg, Pennsylvania
  - Cancer Treatment Centers of America-Eastern Regional Medical Center ( Site 0053), Philadelphia, Pennsylvania
  - Allegheny General Hospital ( Site 0009), Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Centers ( Site 0041), Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System ( Site 0052), Pittsburgh, Pennsylvania
  - Saint Francis Cancer Center ( Site 0096), Greenville, South Carolina
  - Emily Couric Clinical Cancer Center ( Site 0013), Charlottesville, Virginia
  - Inova Schar Cancer Institute ( Site 0032), Fairfax, Virginia
  - Virginia Cancer Specialists, PC ( Site 0080), Fairfax, Virginia
  - Providence Regional Cancer Partnership ( Site 0065), Everett, Washington
- Argentina (10):
  - Centro de Oncologia e Investigacion Buenos Aires COIBA ( Site 0136), Berazategui, Buenos Aires
  - Hospital Privado de Comunidad. ( Site 0130), Mar del Plata, Buenos Aires
  - Hospital Universitario Austral ( Site 0127), Pilar, Buenos Aires
  - Fundacion Favaloro ( Site 0128), Ciudad de Buenos Aires, Buenos Aires F.D.
  - Sanatorio Britanico ( Site 0125), Rosario, Santa Fe Province
  - Sanatorio Parque ( Site 0135), Rosario, Santa Fe Province
  - Hospital Provincial del Centenario ( Site 0131), Rosario, Santa Fe Province
  - Hospital Privado Universitario de Córdoba ( Site 0139), Córdoba
  - Sanatorio Allende ( Site 0129), Córdoba
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica ( Site 0133), San Juan
- Australia (2):
  - Orange Health Services ( Site 0624), Orange, New South Wales
  - Westmead Hospital ( Site 0621), Westmead, New South Wales
- Belgium (6):
  - AZ Sint-Maarten ( Site 0226), Mechelen, Antwerpen
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman ( Site 0223), Liège, Liege
  - UZ Gent ( Site 0224), Ghent, Oost-Vlaanderen
  - AZ Nikolaas ( Site 0225), Sint-Niklaas, Oost-Vlaanderen
  - UZ Leuven ( Site 0221), Leuven, Vlaams-Brabant
  - AZ Delta ( Site 0222), Roeselare, West-Vlaanderen
- Brazil (12):
  - Centro Regional Integrado de Oncologia ( Site 0160), Fortaleza, Ceará
  - Instituto do Cancer do Ceara ( Site 0152), Fortaleza, Ceará
  - Sirio-Libanes Brasilia - Centro de Oncologia - Asa Sul ( Site 0159), Brasília, Federal District
  - Liga Norte Riograndense Contra o Cancer ( Site 0150), Natal, Rio Grande do Norte
  - Hospital de Caridade de Ijui ( Site 0153), Ijuí, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 0146), Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao ( Site 0145), Porto Alegre, Rio Grande do Sul
  - YNOVA Pesquisa Clinica ( Site 0823), Florianópolis, Santa Catarina
  - Fundacao Pio XII - Hospital de Cancer de Barretos ( Site 0144), Barretos, São Paulo
  - Instituto Nacional do Cancer Jose Alencar Gomes da Silva INCA ( Site 0149), Rio de Janeiro
  - Hospital Paulistano - Amil Clinical Research ( Site 0822), São Paulo
  - Hospital Alemao Oswaldo Cruz ( Site 0158), São Paulo
- Canada (5):
  - Princess Margaret Cancer Centre ( Site 0109), Toronto, Ontario
  - CIUSSS du Saguenay-Lac-St-Jean ( Site 0101), Chicoutimi, Quebec
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0110), Montreal, Quebec
  - CIUSSS Ouest de l Ile - St-Mary s Hospital ( Site 0104), Montreal, Quebec
  - McGill University Health Centre ( Site 0111), Montreal, Quebec
- China (15):
  - Tianjin Medical University General Hospital ( Site 0806), Tianjin, Anhui
  - Beijing Cancer Hospital ( Site 0810), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 0811), Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences ( Site 0801), Beijing, Beijing Municipality
  - Peking University Third Hospital ( Site 0812), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 0809), Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Center ( Site 0816), Guangzhou, Guangdong
  - Hunan Cancer Hospital ( Site 0815), Changsha, Hunan
  - Fudan University Shanghai Cancer Center ( Site 0813), Shanghai, Shanghai Municipality
  - Zhongshan Hospital of Fudan University ( Site 0808), Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital-Thoracic Surgery department ( Site 0817), Shanghai, Shanghai Municipality
  - Tang Du Hospital ( Site 0803), Xi’an, Shanxi
  - The First Affiliated Hospital of Zhejiang University ( Site 0804), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital.... ( Site 0814), Hangzhou, Zhejiang
  - Hwa Mei Hospital University of Chinese Academy of Sciences ( Site 0802), Ningbo, Zhejiang
- SA Pohja-Eesti Regionaalhaigla ( Site 1100), Tallinn, Harju, Estonia
- France (11):
  - Hopital Foch ( Site 0243), Suresnes, Ain
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud ( Site 0241), Pierre-Bénite, Auvergne-Rhône-Alpes
  - Nouvel Hopital Civil ( Site 0255), Strasbourg, Bas-Rhin
  - CHU de Toulouse - Hopital Larrey ( Site 0258), Toulouse, Haute-Garonne
  - Clinique Francois Chenieux ( Site 0246), Limoges, Haute-Vienne
  - Centre Hospitalier Metropole Savoie Site de Chambery ( Site 0245), Chambéry, Savoie
  - Centre Hospitalier Annecy Genevois ( Site 0242), Pringy, Savoie
  - CHU de Rouen ( Site 0252), Rouen, Seine-Maritime
  - Hôpital Avicenne - Service d oncologie medicale ( Site 0249), Bobigny, Seine-Saint-Denis
  - H.I.A. Sainte-Anne ( Site 0251), Toulon, Var
  - Institut Curie ( Site 0250), Paris
- Germany (15):
  - Klinikum Esslingen GmbH ( Site 0875), Esslingen am Neckar, Baden-Wurttemberg
  - LKI Lungenfachklinik Immenhausen ( Site 0268), Immenhausen, Hesse
  - Florence Nightingale Krankenhaus ( Site 0874), Düsseldorf, North Rhine-Westphalia
  - Lungenklinik Hemer ( Site 0269), Hemer, North Rhine-Westphalia
  - Mathias Spital Rheine ( Site 0261), Rheine, North Rhine-Westphalia
  - Katholisches Klinikum Koblenz Haus Marienhof ( Site 0873), Koblenz, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus ( Site 0273), Dresden, Saxony
  - Universitaetsklinikum Leipzig AOeR ( Site 0277), Leipzig, Saxony
  - LungenClinic Grosshansdorf GmbH ( Site 0267), Großhansdorf, Schleswig-Holstein
  - Universitaetsklinikum Schleswig Holstein ( Site 0871), Kiel, Schleswig-Holstein
  - Zentralklinik Bad Berka GmbH ( Site 0264), Bad Berka, Thuringia
  - SRH Waldklinikum Gera GmbH ( Site 0272), Gera, Thuringia
  - Evangelische Lungenklinik Berlin ( Site 0274), Berlin
  - HELIOS Klinikum Emil von Behring ( Site 0280), Berlin
  - Asklepios Klinikum Hamburg ( Site 0271), Hamburg
- Ireland (3):
  - Cork University Hospital ( Site 0452), Wilton, Cork
  - St James Hospital ( Site 0451), Dublin
  - Mid Western Cancer Centre ( Site 0450), Limerick
- Italy (10):
  - Istituto Nazionale Tumori ( Site 0309), Milano, Abruzzo
  - Azienda Ospedaliera dei Colli V. Monaldi ( Site 0301), Napoli, Campania
  - IRST-Istituto Scientifico Romagnolo per lo Studio e la cura dei Tumori ( Site 0300), Meldola, Forli-Cesena
  - Istituto Clinico Humanitas Research Hospital ( Site 0314), Rozzano, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda-Oncologia Falck ( Site 0315), Milan, Milano
  - Azienda Ospedaliera San Gerardo ( Site 0308), Monza, Monza E Brianza
  - AOU San Luigi Gonzaga di Orbassano ( Site 0313), Orbassano, Torino
  - Azienda Ospedaliera Spedali Civili di Brescia ( Site 0307), Brescia
  - IRCCS Ospedale San Raffaele di Milano ( Site 0303), Milan
  - Azienda Ospedaliera San Camillo Forlanini ( Site 0311), Roma
- Japan (12):
  - Aichi Cancer Center Hospital ( Site 0765), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0761), Kashiwa, Chiba
  - HP of the Univ. of Occupational and Environmental Health, Japan ( Site 0770), Kitakyushu, Fukuoka
  - Hyogo Cancer Center ( Site 0764), Akashi, Hyōgo
  - St. Marianna University School of Medicine Hospital ( Site 0769), Kawasaki, Kanagawa
  - Kanagawa Cancer Center ( Site 0763), Yokohama, Kanagawa
  - Oita University Hospital ( Site 0766), Yufu, Oita Prefecture
  - Fukushima Medical University Hospital ( Site 0772), Fukushima
  - Hiroshima University Hospital ( Site 0762), Hiroshima
  - National Cancer Center Hospital ( Site 0767), Tokyo
  - Juntendo University Hospital ( Site 0768), Tokyo
  - Tokyo Medical University Hospital ( Site 0771), Tokyo
- Latvia (2):
  - Pauls Stradins Clinical University Hospital ( Site 0911), Riga
  - Riga East Clinical University Hospital ( Site 0912), Riga
- Lithuania (2):
  - LSMUL Kauno Klinikos ( Site 0932), Kaunas
  - Nacionalinis Vezio Institutas ( Site 0931), Vilnius
- Malaysia (2):
  - Sarawak General Hospital ( Site 0782), Kuching, Sarawak
  - University Malaya Medical Centre ( Site 0781), Kuala Lumpur
- Poland (6):
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii ( Site 0487), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka ( Site 0488), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Pulmonologii i Torakochirurgii w Bystrej ( Site 0484), Bystra, Lower Silesian Voivodeship
  - Dolnoslaskie Centrum Onkologii. ( Site 0491), Wroclaw, Lower Silesian Voivodeship
  - Szpital Specjalistyczny w Prabutach Sp. z o.o. ( Site 0483), Prabuty, Pomeranian Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi ( Site 0493), Lodz, Łódź Voivodeship
- Romania (13):
  - S C Pelican Impex SRL ( Site 0506), Oradea, Bihor County
  - Centrul Medical Medicover Victoria ( Site 0514), Bucharest, București
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 0501), Cluj-Napoca, Cluj
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 0515), Cluj-Napoca, Cluj
  - SC Radiotherapy Center Cluj SRL ( Site 0509), Comuna Floresti, Cluj
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 0504), Craiova, Dolj
  - S.C.R.T.C.Radiology Therapeutic Center SRL ( Site 0511), Otopeni, Ilfov
  - S C Oncocenter Oncologie Medicala S R L ( Site 0505), Timișoara, Timiș County
  - Spitalul Sf. Constantin ( Site 0512), Brasov
  - Euroclinic Hospital Bucharest ( Site 0510), Bucharest
  - S.C.Focus Lab Plus S.R.L ( Site 0513), Bucharest
  - Spitalul clinic Judetean de urgenta Constanta ( Site 0508), Constanța
  - Spitalul Judetean de Urgenta .Sf. Ioan cel Nou. ( Site 0503), Suceava
- Russia (9):
  - Chelyabinsk Regional Clinical Oncological Dispensary ( Site 0530), Chelyabinsk, Chelyabinsk Oblast
  - N.N. Blokhin NMRCO ( Site 0521), Moscow, Moscow
  - National Medical Research Radiology Centre ( Site 0535), Moscow, Moscow
  - Medical Rehabilitation Center ( Site 0534), Moscow, Moscow
  - SBHI Leningrad Regional Clinical Hospital ( Site 0524), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 0533), Saint Petersburg, Sankt-Peterburg
  - Municipal Clinical Oncology Center ( Site 0523), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 0529), Kazan', Tatarstan, Respublika
  - Tomsk Scientific Research Institute of Oncology ( Site 0526), Tomsk, Tomsk Oblast
- South Africa (4):
  - Wits Clinical Research ( Site 0570), Parktown-Johannesburg, Gauteng
  - Wilgers Oncology Centre ( Site 0573), Pretoria, Gauteng
  - The Oncology Centre ( Site 0571), Durban, KwaZulu-Natal
  - Cape Town Oncology Trials Pty Ltd ( Site 0572), Kraaifontein, Western Cape
- South Korea (5):
  - National Cancer Center ( Site 0702), Gyeonggi-do, Kyonggi-do
  - The Catholic University of Korea St. Vincent s Hospital ( Site 0705), Gyeonggi-do, Kyonggi-do
  - Asan Medical Center ( Site 0701), Seoul
  - Samsung Medical Center ( Site 0704), Seoul
  - SMG-SNU Boramae Medical Center ( Site 0707), Seoul
- Spain (8):
  - Hospital Germans Trias i Pujol. ICO de Badalona ( Site 0381), Badalona, Barcelona
  - Instituto Catalan de Oncologia - ICO ( Site 0388), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Girona Doctor Josep Trueta ( Site 0386), Girona, La Coruna
  - Hospital Universitario Insular de Gran Canaria ( Site 0383), Las Palmas de Gran Canaria, Las Palmas
  - Hospital de la Santa Creu i Sant Pau ( Site 0385), Barcelona
  - Hospital Universitari Vall d Hebron ( Site 0389), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 0382), Madrid
  - Hospital Virgen del Rocio ( Site 0387), Seville
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital ( Site 0725), Kaohsiung City
  - China Medical University Hospital ( Site 0724), Taichung
  - National Taiwan University Hospital ( Site 0721), Taipei
  - Taipei Veterans General Hospital ( Site 0722), Taipei
  - Tri-Service General Hospital ( Site 0726), Taipei
  - Chang Gung Medical Foundation.Linkou Branch ( Site 0723), Taoyuan District
- Ukraine (9):
  - Cherkassy Regional Oncological Center ( Site 0613), Cherkasy, Cherkasy Oblast
  - City Clinical Hosp.4 of DCC ( Site 0607), Dnipro, Dnipropetrovsk Oblast
  - MI Precarpathian Clinical Oncology Center ( Site 0603), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - MI KhRC Kherson Regional Oncology Dispensary ( Site 0614), Kherson, Kherson Oblast
  - PP PPC Acinus Medical and Diagnostic Centre ( Site 0609), Kropyvnytsky, Kirovohrad Oblast
  - National Cancer Institute of the MoH of Ukraine ( Site 0605), Kyiv, Kyivska Oblast
  - Kyiv City Clinical Oncological Center ( Site 0601), Kyiv, Kyivska Oblast
  - MI Odessa Regional Oncological Centre ( Site 0608), Odesa, Odesa Oblast
  - Zaporizhzhya Regional Clinical Oncology Center ( Site 0606), Zaporizhzhya, Zaporizhzhia Oblast
- United Kingdom (8):
  - Leicester Royal Infirmary ( Site 0447), Leicester, Leicestershire
  - The Clatterbridge Cancer Centre NHS Foundation Trust ( Site 0456), Metropolitan Borough of Wirral, Liverpool
  - Royal Marsden NHS Foundation Trust ( Site 0458), London, London, City of
  - Royal Marsden Hospital ( Site 0457), Sutton, London, City of
  - Nottingham City Hospital Campus ( Site 0441), Nottingham, Nottinghamshire
  - Heartlands Hospital in Birmingham ( Site 0455), Birmingham
  - Freeman Hospital ( Site 0444), Newcastle upon Tyne
  - Plymouth Hospitals NHS Trust ( Site 0443), Plymouth

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Spicer JD, Garassino MC, Wakelee H, Liberman M, Kato T, Tsuboi M, Lee SH, Chen KN, Dooms C, Majem M, Eigendorff E, Martinengo GL, Bylicki O, Rodriguez-Abreu D, Chaft JE, Novello S, Yang J, Arunachalam A, Keller SM, Samkari A, Gao S; KEYNOTE-671 Investigators. Neoadjuvant pembrolizumab plus chemotherapy followed by adjuvant pembrolizumab compared with neoadjuvant chemotherapy alone in patients with early-stage non-small-cell lung cancer (KEYNOTE-671): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2024 Sep 28;404(10459):1240-1252. doi: 10.1016/S0140-6736(24)01756-2. Epub 2024 Sep 14. PMID 39288781
- [Result] Wakelee H, Liberman M, Kato T, Tsuboi M, Lee SH, Gao S, Chen KN, Dooms C, Majem M, Eigendorff E, Martinengo GL, Bylicki O, Rodriguez-Abreu D, Chaft JE, Novello S, Yang J, Keller SM, Samkari A, Spicer JD; KEYNOTE-671 Investigators. Perioperative Pembrolizumab for Early-Stage Non-Small-Cell Lung Cancer. N Engl J Med. 2023 Aug 10;389(6):491-503. doi: 10.1056/NEJMoa2302983. Epub 2023 Jun 3. PMID 37272513
- [Derived] Aredo JV, Wakelee HA. Top advances of the year: Perioperative therapy for lung cancer. Cancer. 2024 Sep 1;130(17):2897-2903. doi: 10.1002/cncr.35357. Epub 2024 May 8. PMID 38717993
- [Derived] Romero Roman A, Campo-Canaveral de la Cruz JL, Macia I, Escobar Campuzano I, Figueroa Almanzar S, Delgado Roel M, Galvez Munoz C, Garcia Fontan EM, Muguruza Trueba I, Romero Vielva L, Cano Garcia JR, Martinez Tellez E, Partida Gonzalez C, Jimenez Lopez MF, Jimenez Maestre U, Mongil Poce R, Sanchez Lorente D, Alvarez Kindelan A, Provencio Pulla M. Outcomes of surgical resection after neoadjuvant chemoimmunotherapy in locally advanced stage IIIA non-small-cell lung cancer. Eur J Cardiothorac Surg. 2021 Jul 14;60(1):81-88. doi: 10.1093/ejcts/ezab007. PMID 33661301
- See also: Merck Clinical Trials Information — http://merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26238&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with resectable stage II, IIIA, and resectable IIIB (T3-4N2) non-small cell lung cancer (NSCLC) were recruited to evaluate the efficacy and safety of pembrolizumab (MK-3475) in combination with platinum doublet neoadjuvant chemotherapy (NAC) before surgery [neoadjuvant phase], followed by pembrolizumab alone after surgery [adjuvant phase].
Pre-assignment Details: Of the 797 participants that were randomized to trial, 795 received treatment. At the time of the primary analysis data cut-off, 523 participants are ongoing in the study.
Period: Overall Study
Arm/Group | NAC + Neoadjuvant/Adjuvant Pembrolizumab | NAC + Neoadjuvant/Adjuvant Placebo
Started | 397 | 400
Treated | 396 | 399
Completed | 0 | 0
Not Completed | 397 | 400
Not completed — Withdrawal by Subject | 10 | 12
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 109 | 141
Not completed — Ongoing in study | 276 | 247

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NAC + Neoadjuvant/Adjuvant Pembrolizumab | NAC + Neoadjuvant/Adjuvant Placebo | Total
Number analyzed (Participants) | 397 | 400 | 797
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (8.5) | 63.6 (8.1) | 63.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 116 | 234
  Male | 279 | 284 | 563
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 34 | 70
  Not Hispanic or Latino | 329 | 333 | 662
  Unknown or Not Reported | 32 | 33 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 124 | 125 | 249
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 250 | 239 | 489
  More than one race | 3 | 10 | 13
  Unknown or Not Reported | 13 | 16 | 29
Histology [Count of Participants; unit: Participants] — Participants were classified according to tumor histology: Squamous or Non-squamous.
  Participants
    Squamous | 171 | 173 | 344
    Non-Squamous | 226 | 227 | 453
Overall Cancer Staging [Count of Participants; unit: Participants] — Participants were categorized by NSCLC stage: Stage II or Stage III. The lower the lung cancer stage, the less the cancer has spread. NSCLC stages can range from I to IV.
  Participants
    Stage II | 118 | 121 | 239
    Stage III | 279 | 279 | 558
PD-L1 Expression Level (50% cutoff) [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression status by immunohistochemistry assay using tumor tissue from an archival or newly obtained biopsy. Participants with a tumor proportion score (TPS) were classified as follows: ≥50% = PD-L1 strongly positive; 1-49% = PD-L1 weakly positive; and <1% = PD-L1 negative.
  Participants
    TPS>=50% | 132 | 134 | 266
    TPS<50% | 265 | 266 | 531
Region [Count of Participants; unit: Participants] — Participants were categorized according to geographic region of site: Non-East Asia and East Asia.
  Participants
    East-Asia | 123 | 121 | 244
    Non-East Asia | 274 | 279 | 553

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival (EFS)
Description: EFS is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause. EFS determined either by biopsy assessed by local pathologist or by investigator-assessed imaging using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1). The EFS for all participants is presented (through database cut-off date of 10-Jul-2023).
Time Frame: Up to approximately 5 years
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NAC + Neoadjuvant/Adjuvant Pembrolizumab | NAC + Neoadjuvant/Adjuvant Placebo
Number analyzed (Participants) | 397 | 400
Months | 47.2 [32.9 to NA] — NA = Upper limit not reached at time of data cut-off | 18.3 [14.8 to 22.1]
Statistical Analysis 1: Comparison: NAC + Neoadjuvant/Adjuvant Pembrolizumab vs NAC + Neoadjuvant/Adjuvant Placebo; Test type: Superiority; p < 0.00001, Log Rank — One-sided p-value based on log-rank test stratified by Stage (II versus III), TPS (>=50% versus <50%), Histology (Squamous versus Non-squamous) and Region (East-Asia versus non-East Asia); Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.48 to 0.72] — Stratified Cox model with Efron's tie handling method with treatment as a covariate stratified by Stage (II versus III), TPS (>=50% versus <50%), Histology (Squamous versus Non-squamous) and Region (East-Asia versus non-East Asia)

2. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization until death from any cause. The OS for all participants is presented (through database cut-off date of 10-Jul-2023).
Time Frame: Up to approximately 5 years
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NAC + Neoadjuvant/Adjuvant Pembrolizumab | NAC + Neoadjuvant/Adjuvant Placebo
Number analyzed (Participants) | 397 | 400
Months | NA [NA to NA] — NA= Median OS, lower limit, and upper limit not reached at time of data cut off | 52.4 [45.7 to NA] — NA= Upper limit not reached at time of data cut off
Statistical Analysis 1: Comparison: NAC + Neoadjuvant/Adjuvant Pembrolizumab vs NAC + Neoadjuvant/Adjuvant Placebo; Test type: Superiority; p = 0.00517, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.56 to 0.93] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Major Pathological Response (mPR) Rate
Description: mPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes following completion of neoadjuvant therapy. The mPR rates as assessed by blinded independent pathologist are presented.
Time Frame: Up to approximately 8 weeks following completion of neoadjuvant treatment (up to Study Week 20)
Population: The analysis population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | NAC + Neoadjuvant/Adjuvant Pembrolizumab | NAC + Neoadjuvant/Adjuvant Placebo
Number analyzed (Participants) | 397 | 400
Percentage of Participants | 30.2 [25.7 to 35.0] | 11.0 [8.1 to 14.5]
Statistical Analysis 1: Comparison: NAC + Neoadjuvant/Adjuvant Pembrolizumab vs NAC + Neoadjuvant/Adjuvant Placebo; Test type: Other — Based on Miettinen & Nurminen method stratified by Stage (II versus III), TPS (>=50% versus <50%), Histology (Squamous versus Non-squamous) and Region (East-Asia versus non-East Asia); p < 0.00001, Stratified Miettinen and Nurminen; Difference in Percentage = 19.2, 95% CI 2-sided [13.9 to 24.7]

4. Secondary Outcome: Pathological Complete Response (pCR) Rate
Description: pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy. The pCR rates as assessed by blinded independent pathologist are presented.
Time Frame: Up to approximately 8 weeks following completion of neoadjuvant treatment (up to Study Week 20)
Population: The analysis population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | NAC + Neoadjuvant/Adjuvant Pembrolizumab | NAC + Neoadjuvant/Adjuvant Placebo
Number analyzed (Participants) | 397 | 400
Percentage of Participants | 18.1 [14.5 to 22.3] | 4.0 [2.3 to 6.4]
Statistical Analysis 1: Comparison: NAC + Neoadjuvant/Adjuvant Pembrolizumab vs NAC + Neoadjuvant/Adjuvant Placebo; Test type: Other — [test comment as in outcome 3, analysis 1]; p < 0.00001, Stratified Miettinen and Nurminen; Difference in Pertentage = 14.2, 95% CI 2-sided [10.1 to 18.7]

5. Secondary Outcome: Change From Baseline in Neoadjuvant Phase in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (Item 29) Score
Description: Change from baseline in GHS/QoL score using the EORTC QLQ-C30 will be determined. The EORTC QLQ-C30 is the most widely used cancer-specific, health-related QoL instrument comprised of 30 individual items arranged as both multi-item scales and individual items. Specifically, these items are divided into 5 functional scales (15 items total), 3 symptom scales (7 items total), 6 individual items, and a GHS/QoL scale composed of 2 items: GHS and QoL. The GHS/QoL score measured here refers to only the composite score calculated for the GHS/QoL scale. Both items on the GHS/QoL scale are scored from 1 (very poor GHS/QoL) to 7 (excellent GHS/QoL) and scores for both items are averaged and a linear transformation applied to standardize the overall GHS/QoL score from 0 to 100, with higher overall scores indicating higher GHS/QoL.
Time Frame: Baseline (cycle 1 in neoadjuvant phase) and neoadjuvant week 11
Population: All randomized participants who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Item 30 assessment data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Sore on a scale
Arm/Group | NAC + Neoadjuvant/Adjuvant Pembrolizumab | NAC + Neoadjuvant/Adjuvant Placebo
Number analyzed (Participants) | 390 | 395
Sore on a scale | -9.31 [-11.67 to -6.94] | -10.73 [-13.07 to -8.40]
Statistical Analysis 1: Comparison: NAC + Neoadjuvant/Adjuvant Pembrolizumab vs NAC + Neoadjuvant/Adjuvant Placebo; Test type: Other — Based on a constrained longitudinal data analysis (cLDA) model with the scores as the response variable with covariates for treatment by visit interaction and stratification factors (Stage (II versus III), TPS (>=50% versus <50%), Histology (Squamous versus Non-squamous) and Region (East-Asia versus non-East Asia); p = 0.3611, t-test, 2 sided; Difference in Least Square Means = 1.43, 95% CI 2-sided [-1.64 to 4.49]

6. Secondary Outcome: Change From Baseline in Adjuvant Phase in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (Item 29) Score
Description: as for outcome 5
Time Frame: Baseline (cycle 1 in neoadjuvant phase) and adjuvant week 10 (up to Study Week 30)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Sore on a scale
Arm/Group | NAC + Neoadjuvant/Adjuvant Pembrolizumab | NAC + Neoadjuvant/Adjuvant Placebo
Number analyzed (Participants) | 395 | 397
Sore on a scale | -1.52 [-3.67 to 0.63] | -3.74 [-5.96 to -1.52]
Statistical Analysis 1: Comparison: NAC + Neoadjuvant/Adjuvant Pembrolizumab vs NAC + Neoadjuvant/Adjuvant Placebo; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.1197, t-test, 2 sided; Difference in Least Square Means = 2.22, 95% CI 2-sided [-0.58 to 5.02]

7. Secondary Outcome: Number of Participants Who Experience an Adverse Event (AE)
Time Frame: Up to approximately 71 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

8. Secondary Outcome: Number of Participants Who Experience Perioperative Complications
Description: Perioperative complications are a discrete set of both intraoperative and postoperative complications, potentially contributing to increased length of inpatient care and/or delay of adjuvant therapy. The number of participants experiencing perioperative complications will be assessed.
Time Frame: Up to approximately 51 weeks following surgery
Population: The analysis population consisted of all randomized participants who received at least one dose of neoadjuvant study treatment and also undergo on-study surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | NAC + Neoadjuvant/Adjuvant Pembrolizumab | NAC + Neoadjuvant/Adjuvant Placebo
Number analyzed (Participants) | 325 | 317
Participants | 233 | 229

9. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Time Frame: Up to approximately 57 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

ADVERSE EVENTS:
Time Frame: Up to approximately 71 weeks
Description: All-Cause Mortality includes all randomized participants. Serious and Other adverse events (AEs) includes all randomized participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs.
Groups:
- Pembro + Chemo/Pembro: Neoadjuvant: Prior to surgery, participants receive up to 4 cycles (cycle length: 3 weeks) of pembrolizumab [200 mg, intravenous (IV); given on cycle day 1] in combination with platinum doublet neoadjuvant chemotherapy (NAC), consisting of cisplatin [75 mg/m^2, IV; given on cycle day 1] and either Gemcitabine [1000 mg/m^2, IV; given on cycle days 1 and 8] or Pemetrexed [500 mg/m^2, IV; given on cycle day 1].
  Adjuvant: 4-12 weeks following surgery, participants receive 13 cycles (cycle length: 3 weeks) of pembrolizumab [200 mg, IV; given on cycle day 1].
- Placebo + Chemo/Placebo: Neoadjuvant: Prior to surgery, participants receive up to 4 cycles (cycle length: 3 weeks) of placebo [normal saline, IV; given on cycle day 1] in combination with platinum doublet NAC, consisting of cisplatin [75 mg/m^2, IV; given on cycle day 1] and either Gemcitabine [1000 mg/m^2, IV; given on cycle days 1 and 8] or Pemetrexed [500 mg/m^2, IV; given on cycle day 1].
  Adjuvant: 4-12 weeks following surgery, participants receive 13 cycles (cycle length: 3 weeks) of placebo [normal saline, IV; given on cycle day 1].
Arm/Group | Pembro + Chemo/Pembro | Placebo + Chemo/Placebo
All-Cause Mortality (participants affected / at risk) | 110/397 | 144/400
Serious Adverse Events (participants affected / at risk) | 165/396 | 133/399
Other Adverse Events (participants affected / at risk) | 389/396 | 388/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembro + Chemo/Pembro (N=396) | Placebo + Chemo/Placebo (N=399)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 3 (4)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 3 (3)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 3 (3)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (2)
General physical health deterioration (General disorders) | 3 (4) | 1 (1)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 8 (8) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 21 (25) | 19 (21)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Systemic infection (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Anastomotic fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Epidural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (6) | 1 (1)
Platelet count decreased (Investigations) | 3 (3) | 10 (10)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenic syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 3 (3)
Renal impairment (Renal and urinary disorders) | 1 (1) | 3 (3)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (7)
Pleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (9)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembro + Chemo/Pembro (N=396) | Placebo + Chemo/Placebo (N=399)
Anaemia (Blood and lymphatic system disorders) | 163 (229) | 165 (233)
Tinnitus (Ear and labyrinth disorders) | 29 (31) | 23 (25)
Hypothyroidism (Endocrine disorders) | 42 (46) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 22 (22) | 18 (19)
Constipation (Gastrointestinal disorders) | 154 (207) | 146 (205)
Diarrhoea (Gastrointestinal disorders) | 78 (113) | 73 (101)
Dyspepsia (Gastrointestinal disorders) | 24 (28) | 22 (26)
Nausea (Gastrointestinal disorders) | 228 (385) | 210 (347)
Stomatitis (Gastrointestinal disorders) | 41 (52) | 36 (42)
Vomiting (Gastrointestinal disorders) | 81 (119) | 68 (103)
Asthenia (General disorders) | 58 (73) | 65 (95)
Chest pain (General disorders) | 46 (48) | 33 (37)
Fatigue (General disorders) | 125 (174) | 101 (139)
Malaise (General disorders) | 36 (46) | 28 (49)
Oedema peripheral (General disorders) | 40 (47) | 24 (29)
Pyrexia (General disorders) | 43 (55) | 31 (33)
Pneumonia (Infections and infestations) | 15 (17) | 20 (22)
Upper respiratory tract infection (Infections and infestations) | 21 (22) | 12 (18)
Urinary tract infection (Infections and infestations) | 20 (25) | 16 (23)
Incision site pain (Injury, poisoning and procedural complications) | 23 (23) | 18 (18)
Procedural pain (Injury, poisoning and procedural complications) | 61 (62) | 59 (59)
Alanine aminotransferase increased (Investigations) | 57 (81) | 40 (64)
Aspartate aminotransferase increased (Investigations) | 42 (63) | 32 (45)
Blood creatinine increased (Investigations) | 69 (101) | 59 (88)
Blood urea increased (Investigations) | 21 (32) | 16 (22)
Lymphocyte count decreased (Investigations) | 24 (46) | 26 (56)
Neutrophil count decreased (Investigations) | 171 (296) | 169 (303)
Platelet count decreased (Investigations) | 74 (115) | 73 (106)
Weight decreased (Investigations) | 32 (35) | 24 (26)
White blood cell count decreased (Investigations) | 112 (202) | 102 (202)
Decreased appetite (Metabolism and nutrition disorders) | 115 (166) | 102 (147)
Hyperglycaemia (Metabolism and nutrition disorders) | 26 (49) | 42 (68)
Hyperkalaemia (Metabolism and nutrition disorders) | 32 (48) | 20 (31)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 19 (32) | 23 (41)
Hypokalaemia (Metabolism and nutrition disorders) | 30 (48) | 40 (51)
Hypomagnesaemia (Metabolism and nutrition disorders) | 49 (70) | 41 (72)
Hyponatraemia (Metabolism and nutrition disorders) | 41 (79) | 36 (74)
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 (42) | 35 (44)
Back pain (Musculoskeletal and connective tissue disorders) | 36 (44) | 24 (29)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 (22) | 10 (12)
Dizziness (Nervous system disorders) | 51 (62) | 45 (56)
Dysgeusia (Nervous system disorders) | 31 (35) | 36 (36)
Headache (Nervous system disorders) | 43 (50) | 41 (45)
Insomnia (Psychiatric disorders) | 51 (57) | 26 (31)
Cough (Respiratory, thoracic and mediastinal disorders) | 74 (91) | 60 (63)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 71 (79) | 51 (54)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 27 (36) | 36 (46)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 27 (27)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 26 (28)
Alopecia (Skin and subcutaneous tissue disorders) | 45 (45) | 41 (41)
Pruritus (Skin and subcutaneous tissue disorders) | 53 (56) | 35 (37)
Rash (Skin and subcutaneous tissue disorders) | 69 (85) | 34 (47)
Hypertension (Vascular disorders) | 34 (44) | 38 (41)
Hypotension (Vascular disorders) | 20 (21) | 15 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT03425643/Prot_SAP_000.pdf